CLINICAL TRIAL: NCT00713648
Title: A Multi-Centre, Open-Label, Single-Arm and Multiple Dosing Trial on Efficacy and Safety of Monthly Replacement Therapy With Recombinant Factor XIII (rFXIII) in Subjects With Congenital Factor XIII Deficiency
Brief Title: Evaluation of Recombinant Factor XIII for Prevention of Bleeding in Patients With FXIII Inherited Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F13CD-1725; 2006-003148-51 (EudraCT Number)
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — 35 IU/kg body weight, i.v. administration, once every 4 weeks

SUMMARY:
The trial is conducted in Europe, North America and Asia. The aim of this trial is to evaluate catridecacog (recombinant factor XIII (rFXIII)) treatment in patients with inherited FXIII deficiency. It is expected that recombinant FXIII can be used for the prevention of bleeding episodes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital FXIII A-subunit deficiency (confirmed by genotyping at screening visit)
* Treatment with regular FXIII replacement therapy initiated at least 6 months prior to screening and one of the following : a documented history of at least one 1 treatment-requiring bleeding episode prior to initiation of regular replacement therapy or a documented family history of FXIII congenital deficiency (only for subjects on regular replacement therapy prior to screening)
* Documented history of at least two 2 bleeding episodes requiring treatment with FXIII containing blood products within the last 12 months prior to screening (only for subjects receiving on-demand treatment prior to screening)

Exclusion Criteria:

* Known neutralizing antibodies (inhibitors) towards FXIII
* Any known congenital or acquired coagulation disorder other than congenital FXIII deficiency
* Documented history of at least 2 treatment-requiring bleeding episodes per year during previous regular replacement therapy with FXIII containing blood products (fresh frozen plasma (FFP), plasma-derived FXIII (pd FXIII) and cryoprecipitate)
* Known or suspected allergy to trial product(s) or related products
* Planned major surgery during the trial period. Catheter, ports and dental extractions do not count as surgeries and will not exclude the subject
* Renal insufficiency defined as current dialysis therapy
* Any history of confirmed venous or arterial thrombo-embolic events

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- United States (11):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Seattle, Washington
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Klagenfurt
  - Novo Nordisk Investigational Site, Vienna
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (3):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
- Germany (3):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Braunschweig
  - Novo Nordisk Investigational Site, Duisburg
- Israel (2):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Vicenza, Italy
- Spain (2):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Seville
- Novo Nordisk Investigational Site, Zurich, Switzerland
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Result] Inbal A, Oldenburg J, Carcao M, Rosholm A, Tehranchi R, Nugent D. Recombinant factor XIII: a safe and novel treatment for congenital factor XIII deficiency. Blood. 2012 May 31;119(22):5111-7. doi: 10.1182/blood-2011-10-386045. Epub 2012 Mar 26. PMID 22451421
- [Result] Brand-Staufer B, Carcao M, Kerlin BA, Will A, Williams M, Tornoe CW, Sandberg Lundblad M, Nugent D. Pharmacokinetic characterization of recombinant factor XIII (FXIII)-A2 across age groups in patients with FXIII A-subunit congenital deficiency. Haemophilia. 2015 May;21(3):380-385. doi: 10.1111/hae.12616. Epub 2015 Jan 21. PMID 25643920
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of a total of 29 initiated trial sites, 23 sites enrolled and dosed at least one patient. The country distribution was (number of actively recruiting sites per country in parenthesis): Austria (1), Canada (1), Finland (1), France (1), Germany (3), Israel (2), Italy (1), Spain (1), Switzerland (1), UK (3) and United States of America (8)
Pre-assignment Details: After screening, eligible subjects entered a 4-week run-in period followed by a 52-week recombinant factor XIII (rFXIII) treatment period. Subjects who before entering the trial were receiving regular replacement therapy with a FXIII-containing product were to receive their last standard replacement dose just before the screening visit.
Groups:
- rFXIII: Subjects received 35 IU/kg rFXIII every 4th week (28±2 days) during a treatment period of 52 weeks. In case of acute bleeding episodes, any additional treatment as per investigator judgment was to be according to local standard practice. Additional doses of rFXIII could therefore not be used to treat such breakthrough bleedings
Period: Overall Study
Arm/Group | rFXIII
Started | 41
Completed | 33
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Unclassified | 2
Not completed — According to Protocol | 2
Not completed — Development of antibodies | 3

BASELINE CHARACTERISTICS:
Arm/Group | rFXIII
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (15.9)
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2
  White | 28
  Asian | 5
  Other | 5
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate (Number Per Subject Year) of Bleeding Episodes Requiring Treatment With a FXIII Containing Product During the Treatment Period
Description: It represents the incidence of bleeding episodes requiring treatment with a FXIII-containing product.
Time Frame: For a period of 322 days (approximately one year) comprised of a screening visit (Visit 1), treatment period (Visits 2-15), unscheduled visit and end-of-trial visit (Visit 16).
Population: Full analysis set - consisting of a total of 41 subjects who received at least one dose of trial product.
Measure: Mean (Full Range); unit: bleeding episodes per subject per year
Arm/Group | rFXIII
Number analyzed (Participants) | 41
bleeding episodes per subject per year | 0.138 [0 to 2]
Statistical Analysis 1: Comparison: rFXIII; Test type: Superiority or Other; Poisson model (log-link); The estimated rate was adjusted for age and overdispersion which was estimated by Pearson's chi-square statistic divided by its degrees of freedom; Mean (Lambda) = 0.048, 95% CI [0.0094 to 0.2501] — Mean (Lambda) refer to the estimate of the annualised bleeding rate

2. Secondary Outcome: Percentage of Subjects Having a Normal Clot Solubility One Hour After rFXIII Administration and 28 Days After rFXIII Administration for All Dosing Visits
Description: Blood samples for clot solubility drawn at each visit (1 hour before and after dose administration). A clot solubility assay was used to screen for FXIII deficiency. The assay is based on the ability of urea to dissolve fibrin clots that have not undergone FXIII-induced stabilization. Normal blood clots generally remain stable for 24 hours or more, while clots in which fibrin molecules have not been cross-linked are soluble within minutes. The outcome of the test is normal (FXIII present; a clot is observed in the test tube) or abnormal (FXIII absent or very low level; no clot in test tube).
Time Frame: as for outcome 1
Population: Full analysis set - consisting of a total of 41 subjects who received at least one dose of trial product. For All Dosing Visits, the participants analyzed (N) are the 'All Visit Subjects Count' i.e. the sum of subject counts across all dosing visits combined.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | rFXIII
Number analyzed (Participants) | 41
percentage (%) of subjects
  After 1 hour post-dosing (N=444) | 98.2
  After 28 days of treatment (N=419) | 91.3

3. Secondary Outcome: Level of FXIII Activity One Hour After rFXIII Administration and 28 Days After rFXIII Administration for All Dosing Visits
Description: Subjects entered a 52-week treatment period of monthly (28±2 days) doses of 35 IU/kg rFXIII. Blood samples for analysis of FXIII activity were drawn at each visit; at dosing visits blood was drawn 1 hour after administration and before administration(corresponding to 28 days after the previous dose). All Dosing Visits are visits where a dose is given (i.e. Visit 2-15 except Visit 3).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | rFXIII
Number analyzed (Participants) | 41
U/kg
  After 1 hour post-dosing (N=453) | 0.782 (0.342)
  After 28 days of treatment (N=459) | 0.189 (0.102)

4. Secondary Outcome: Number of Subjects With rFXIII Antibody Development
Description: Subjects receiving rFXIII were monitored for the development of binding antibodies. Blood sampling was done before administration of trial product at all visits (Visits 1-16 and unscheduled visit)
Time Frame: as for outcome 1
Population: Full analysis set - Subjects who received at least one dose of trial product.
Measure: Number; unit: participants
Arm/Group | rFXIII
Number analyzed (Participants) | 41
participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected and reported during the entire study period i.e. approximately one year (322 days)
Description: All AEs observed by the investigator or reported spontaneously by the subjects, were recorded by the investigator at each contact with the site (visit or telephone, excluding safety visits, where the subject was not seeing the Investigator or his staff (e.g.visits to the laboratory))
Arm/Group | rFXIII
Serious Adverse Events (participants affected / at risk) | 6/41
Other Adverse Events (participants affected / at risk) | 25/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII (N=41)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Antibody test positive (Investigations) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII (N=41)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 7 (7)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 8 (11)
Urinary tract infection (Infections and infestations) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 3 (3)
Incorrect dose administered (Injury, poisoning and procedural complications) | 4 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 11 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk (NN) reserves the right not to release data until after specified milestones, e.g., finalisation of clinical trial report. This includes the right not to release interim results of clinical trials, as release of such information can invalidate the trial results. At end of trial, one or more manuscripts will be prepared collaboratively between Investigator(s) and NN. NN reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.